CLINICAL TRIAL: NCT03234270
Title: Changes in Aviators' Body Core Temperature Measurements at F-35
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Israeli Air Force Aeromedical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Coretemp 1799-2017
Record Dates: First submitted 2017-07-26; First posted 2017-07-31 (Actual); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Aviation; Heat Stress
Keywords: Heat stress, pilots
MeSH Terms: conditions — Heat Stress Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- F35 pilots (Experimental)
  Interventions: Device: Core temperature measurements
- F15 pilots (Active Comparator)
  Interventions: Device: Core temperature measurements

INTERVENTIONS:
Device: Core temperature measurements — Core temperature measurements with coretemp pill

SUMMARY:
The many complaints that have been expressed by the US aircrew of the F-35 regarding the heat stress in the cockpit raised an obvious concern that, as a result of such heat levels, the aviators' core body temperature may increase significantly, and subsequently cause severe cognitive impairment- risking both the pilot and the mission.

In order to validate this hypothesis, we will measure the aviators' core body temperatures while inside the cockpit of the F-35, to see whether their core body temperatures are rising to a level that can cause heat stress or not. The temperatures will be measured on another fourth generation aircraft as well for comparing purposes.

The temperatures will be measured using a Telemetric pill which will be ingested by each aviator. Once ingested, the pill will transmit the data to an external monitor. The collected data will be examined and analyzed in order to determine the likelihood of heat stress occurrence.

ELIGIBILITY:
Inclusion Criteria:

* F35 pilots
* Signing on informed consent

Exclusion Criteria:

* Sickness two weeks prior the experiment

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-07 (Estimated); Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Mean core temp. of F35 pilots in hot weather conditions | 40 minutes

IPD SHARING:
Plan to Share IPD: No